CLINICAL TRIAL: NCT02130648
Title: Non-invasive Prenatal Diagnosis (NIPD) of Cystic Fibrosis by Quantitative Real Time MEMO-PCR
Brief Title: Non Ivasive Prenatal Diagnosis (NIPD) of Cystic Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: UF9039
Record Dates: First submitted 2014-04-22; First posted 2014-05-05 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-04

CONDITIONS: Noninvasive Mucinous Cystadenocarcinoma of Ovary
Keywords: Non-invasive Prenatal Diagnosis (NIPD); Cystic Fibrosis; Quantitative real time MEMO-PCR
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prenatal diagnosis: Prenatal diagnosis witch A sampling of blood de 14 ml
  Interventions: Other: A sampling of blood

INTERVENTIONS:
Other: A sampling of blood — A sampling of blood de 14 ml

SUMMARY:
The purprose of this study is to develop and validate an analytical and clinical NIPD test for cystic fibrosis from maternal blood by analysis circulating free fetal DNA (cff-DNA), searching for the paternal mutation in families with CFTR compound heterozygosity

DETAILED DESCRIPTION:
The recent development of techniques to analyze foetal DNA circulating in blood maternal opened new perspectives for prenatal diagnosis (PD). Non-invasive PND (NIPD) is now the method of choice for the determination of fetal sex (genetic disorders linked to X chromosome) and rhesus genotype. NIPD begins to find applications in the diagnosis of monogenic diseases for mutations of paternal transmission. However a number of technical challenges still hamper diagnostic applications in routine, and have to be resolved taking into account the aspects of cost, reliability (false negative ..) and complexity of equipment and bioinformatics studies.

The investigators propose to develop and validate an analytical and clinical NIPD test for cystic fibrosis from maternal blood by analysis circulating free fetal DNA (cff-DNA), searching for the paternal mutation in families with CFTR compound heterozygosity.

The test method based on MEMO associated with a platform for real-time PCR can be used for the detection of trace DNA mutant. This technique is commonly used for mutations in mosaic (less than 1%) of genes common cancers. Positive detection of the paternal mutation is always checked by a second mini-sequencing technique.

Prior to any specific CFTR test, the DNA profile of each sample will be determined using a commercial kit of Mini STR adapted to study casework. A tri-allelic profile for markers will prove the presence of fetal DNA in the studied specimen and will thus limit false negatives associated with the lack or insufficient amounts of cff-DNA.

The validation step of the investigators analytical methods will be made on chimeric DNA control samples artificially created. Then the test will be clinicaly validated by a retrospective study of maternal serum from pregnant women, who have been the subject of PND or PGD (preimplantation genetic diagnosis) of CF request in the laboratory during the study period (2012 to 2013).

The investigators structure is a reference center for PGD, PND and NBS (newborn screening) of cystic fibrosis. The samples will be collected in accordance with current regulations.The pre-analytical sample treatment will be done in real time and plasma will be stored for the second step of the study.

The validation of the proposed tests will permit :

* To have an external quality control (QC) confirming the presence of a minor DNA in the studied sample. This QC could be used for all NIPD tests based on the search of a genomic sequence absent from the maternal genome
* To have a highly sensitive method to detect trace mutant DNA which can be develop for new NIPD tests in other monogenic diseases by detecting mutations of the same nature.

The investigators project, limited to the search for the paternal allele in the family with CFTR compound heterozygosity, is a first step in the implementation of a prenatal diagnosis approach of cystic fibrosis that the investigators aim to develop in order to to reduce invasive procedures.

ELIGIBILITY:
Inclusion criteria:

* pregnant women with a risk of cystic fibrosis for the foetus

Exclusion criteria:

* both parents have the same CF mutant allele

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women with a risk of cystic fibrosis for the foetus
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-07 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Analysis circulating free fetal DNA | 10th week with regard to the term of the pregnancy
  Analytical and clinical NIPD test for cystic fibrosis from maternal blood by analysis circulating free fetal DNA (cff-DNA), searching for the paternal mutation in families with CFTR compound heterozygosity.
  The test method based on MEMO associated with a platform for real-time PCR can be used for the detection of trace DNA mutant.

CONTACTS AND LOCATIONS:
Overall Officials: Mireille CLAUSTRES, Principal Investigator — Laboratoire de Genetique Moleculaire Institut de Recherche Clinique INSERM 827 640, avenue du Doyen giraud 34295 MONTPELLIER cedex 5
Locations (1):
- Centre hospitalier Universitaire de Montpellier, Montpellier, France